CLINICAL TRIAL: NCT05279547
Title: Locomotor Muscle Oxygenation and Activation During Acute Interval Compared to Constant-load Bed-cycling Exercise: A Pilot Study
Brief Title: Locomotor Muscle Oxygenation and Activation During Acute Interval Compared to Constant-load Bed-cycling Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Daniel Langer, Prof. Dr, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S65934
Record Dates: First submitted 2022-02-15; First posted 2022-03-15 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Intensive Care Unit Acquired Weakness; Critical Illness
Keywords: ICU acquired muscle weakness; Quadriceps muscle; Near-infrared spectroscopy; Oxygenation; EMG; Early-mobilization; Bed-cycling; Interval exercise; Continuous exercise
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: two arms randomized cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (First constant-load then interval bed-cycling protocol) (Active Comparator): During Day 1, patients will be familiarized with the constant-load and interval bed-cycling exercise against no resistance. Patients will be also randomized in the two arms of the study before the determination of the appropriate exercise intensities to be subsequently use during the constant-load and interval bed-cycling protocols on Day 2 and Day 3. Exercise intensities will be determined so that the volume of training during the two protocols will be equal.
  During Day 2, patients randomized to arm 1 will perform the constant-load bed-cycling protocol. During Day 3, patients who executed the constant-load bed-cycling protocol on Day 1 (arm 1) will perform the interval bed-cycling protocol.
  Interventions: Other: Constant-load bed-cycling exercise; Other: Interval bed-cycling exercise
- Arm 2 (First interval then constant-load bed-cycling protocol) (Active Comparator): During Day 1, patients will be familiarized with the constant-load and interval bed-cycling exercise against no resistance. Patients will be also randomized in the two arms of the study before the determination of the appropriate exercise intensities to be subsequently use during the constant-load and interval bed-cycling protocols on Day 2 and Day 3. Exercise intensities will be determined so that the volume of training during the two protocols will be equal.
  During Day 2, patients randomized to arm 2 will perform the interval bed-cycling protocol. On Day 3 they will perform the constant-load bed-cycling protocol.
  Interventions: Other: Constant-load bed-cycling exercise; Other: Interval bed-cycling exercise

INTERVENTIONS:
Other: Constant-load bed-cycling exercise — Patients will actively cycle for a minimum duration of 10 minutes and a maximum duration of 20 minutes without breaks.
Other: Interval bed-cycling exercise — Patients will cycle for the same duration as during constant-load exercise. Interval bed-cycling session will consist of 30 seconds of high intensity exercise alternated by 30 seconds of passive cycling designed so that volume of training will be equal.

SUMMARY:
Up to 60% of patients admitted to the Intensive Care Unit (ICU) with a prolonged stay in the ICU develop complications such as intensive care unit acquired weakness (ICUAW) characterized by limb and respiratory muscle weakness. ICUAW is associated with worse prognosis, longer ICU stay and increased morbidity and mortality.

Physical therapy (PT) interventions in the intensive care unit (ICU), can improve patients' outcomes.

However, improvements in muscle function achieved with standard physical activity interventions aiming at early mobilization are highly variable due to lack of consistency in definition of the interventions, lack of consideration for the complexity of exercise dose and/or insufficient stimulation of muscles during interventions. It has been suggested that modifying early mobilization and exercise protocols towards shorter intervals consisting of higher intensity exercises might result in more optimal stimulation of muscles.

In the present study the researchers therefore aim to simultaneously assess (by non-invasive technologies) locomotor muscle oxygenation and activation along with the measurements of the load imposed on respiration and circulation during two different training modalities i.e., moderate intensity continuous bed-cycling (endurance training) vs high-intensity alternated by lower intensity periods of bed-cycling (interval training).

DETAILED DESCRIPTION:
Critical illness is related to high morbidity and mortality rates, and health-care costs. Up to 60% of patients admitted to the Intensive Care Unit (ICU) with a prolonged stay in the ICU develop complications such as intensive care unit acquired weakness (ICUAW) characterized by limb and respiratory muscle weakness. These abnormalities develop already within the first days to weeks after intensive care unit (ICU) admission and are related to immobility, sepsis, inflammatory response syndrome (SIRS), prolonged mechanical ventilation, multiple organ failure, and the use of corticosteroids. ICUAW is associated with worse prognosis, longer ICU stay and increased morbidity and mortality. Survivors of critical illness frequently report long-term physical impairments persisting up to 5 years after discharge.

Physical therapy (PT) interventions in the intensive care unit (ICU), can improve patients' outcomes. A systematic review of randomized controlled trials (RCTs) of strategies to improve physical functioning of ICU survivors identified the importance of PT interventions in the ICU. Early rehabilitation during ICU admission has the potential to result in important clinical benefits for patients. These findings highlight the importance of aiming to apply mobilization strategies early during ICU stay to maintain and improve physical functioning as good as possible.

With a projected increase in the number of critically ill patients, requiring rehabilitation in the ICU effective and efficient rehabilitation interventions are warranted. However, improvements in muscle function achieved with standard physical activity interventions aiming at early mobilization are highly variable. Therefore, there is a need for implementing more evidence-based PT interventions, as part of routine clinical practice. Variable results of current interventions may be due to lack of consistency in definition of the interventions, lack of consideration for the complexity of exercise dose and/or insufficient stimulation of muscles during interventions. It has been suggested that modifying early mobilization and exercise protocols towards shorter intervals consisting of higher intensity exercises might result in more optimal stimulation of muscles.

A recent study evaluating a cohort of 181 consecutive patients receiving 541 in-bed cycling sessions as part of routine PT interventions in ICU showed that constant-load bed-cycling appears to be both feasible and safe. In addition, recent evidence in patients with chronic lung disease shows that acute alteration of intense and less intense periods of exercise induced partial restoration of local muscle oxygen stores during the less intense periods of exercise facilitating the muscles to achieve higher exercise intensities during the intense periods, compared to constant-load submaximal exercise. Hence, in patients with chronic lung diseases, alternating intense with less intense loads during interval exercise may be physiologically more effective than constant submaximal workloads maintained during endurance type training for achieving a higher stimulation of locomotor muscles. This has not been investigated so far in intensive care unit patients.

ELIGIBILITY:
Inclusion Criteria:

* Full cooperatively adult patients indicated by the Adequacy Score of standardized 5 questions (SQ5) = 5/5
* Patients mechanically ventilated for longer than 48 hours during the same ICU admission
* Patients are expected to remain in the ICU for more than an additional 48 hours starting from study enrollment
* Patients able to perform active cycling for > 10 consecutive minutes

Exclusion Criteria:

* Pre-existing functional limitations
* Low limb injuries or conditions that would preclude in-bed cycling such as a body habitus unable to fit the bike
* Extreme obesity (body mass index >35 kg/m2)
* Neurologically unstable
* Acute surgery
* Palliative goals of care
* Temperature > 40 °C
* An anticipated fatal outcome
* Evidence of coronary ischaemia, for example, chest pain or electrocardiogram changes
* Resting heart rate <40 or >120 beats per minute
* Mean arterial pressure <60 or >120 mmHg
* Peripheral capillary oxygen saturation < 90%
* Wounds, trauma or surgery of leg precluding cycle ergometry
* Wounds, trauma or surgery of pelvis precluding cycle ergometry
* Wounds, trauma or surgery of lumbar spine precluding cycle ergometry
* Coagulation disorder (international normalised ratio > 1.8, or platelets < 50,000 mcL)
* Intracranial pressure >20 mm Hg
* Femoral access other than femoral central line
* Acute deep vein thrombosis
* Pulmonary embolism
* >20 mcg/min of noradrenaline
* inotropic or vasopressor support comparable to a dose of noradrenaline >20mcg/min
* Fraction of inspired oxygen > 55%
* Arterial partial pressure of oxygen (PaO2) <65 torr (<8.66 kPa)
* Positive end-expiratory pressure > 10 cmH2O
* Respiratory rate > 30 breaths per minutes with adequate ventilatory support
* Minute ventilation >150 mL/kg body weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Differences between bed-cycling protocols in fractional oxygen saturation (StiO2,%) for each measured region of the m. quadriceps femoris | constant-load and interval bed-cycling protocols administered in 2 different days within 1 week
  Assessed by near-infrared spectroscopy
Differences between bed-cycling protocols in activation (sEMG amplitude) for each measured region of the muscle quadriceps femoris | constant-load and interval bed-cycling protocols administered in 2 different days within 1 week
  Assessed by surface electromyography
Adverse event rate during constant-load bed-cycling | 1 session of maximal 20 minutes of constant-load bed-cycling per patient
  Constant-load bed-cycling protocol will be considered as a safe intervention in case the adverse event rate will be less than 2.6%; adverse events: catheter/tube removal, increase in vasoactive medications >5mcg/min, increase in systolic blood pressure > 200 mmHg for > 2min, decrease in mean arterial pressure < 60 mmHg for > 2 min, decrease in heart rate < 50 bpm for > 2 min, increase in heart rate > 140 beats per minute for > 2 min, increase in respiratory rate and sustained > 5 min after session, decrease in peripheral capillary oxygen saturation < 88% for > 1 min requiring an increase in fraction of inspired oxygen > 0.1 sustained > 5 min)
Adverse event rate during interval bed-cycling | 1 session of maximal 20 minutes of interval bed-cycling per patient
  Interval bed-cycling protocol will be considered as a safe intervention in case the adverse event rate will be less than 2.6%; adverse events: catheter/tube removal, increase in vasoactive medications >5mcg/min, increase in systolic blood pressure > 200 mmHg for > 2min, decrease in mean arterial pressure < 60 mmHg for > 2 min, decrease in heart rate < 50 bpm for > 2 min, increase in heart rate > 140 beats per minute for > 2 min, increase in respiratory rate and sustained > 5 min after session, decrease in peripheral capillary oxygen saturation < 88% for > 1 min requiring an increase in fraction of inspired oxygen > 0.1 sustained > 5 min)
Percentage of completed constant-load bed-cycling sessions | 1 session of maximal 20 minutes of constant-load bed-cycling per patient
  The constant-load bed-cycling is deemed to be feasible if at least 80% of planned constant-load sessions were able to be commenced and 80% of commenced sessions can be completed
Percentage of completed interval bed-cycling sessions | 1 session of maximal 20 minutes of interval bed-cycling per patient
  The interval bed-cycling is deemed to be feasible if at least 80% of planned interval sessions were able to be commenced and 80% of commenced sessions can be completed

SECONDARY OUTCOMES:
Differences in Relative dispersion (RD) of fractional oxygen saturation (StiO2,%) among the different regions of quadriceps femoris as indicator of heterogeneity of fractional oxygen extraction among different regions of quadriceps femoris muscle. | 1 session constant-load bed-cycling + 1 interval bed-cycling session administered in 2 different days within 1 week.
  Differences between exercise protocols in Relative dispersion (RD) of fractional oxygen saturation (StiO2,%) among the different regions of quadriceps femoris (i.e., vastus lateralis, vastus medialis, rectus femoris upper part and rectus femoris lower part) as indicator of heterogeneity of fractional oxygen extraction among different regions of quadriceps femoris muscle.
Differences between exercise protocols in oxygenated hemoglobin/myoglobin (OxyHb/Mb), deoxygenated hemoglobin/myoglobin (DeoxyHb/Mb) and total hemoglobin/myoglobin concentration (TotHb/Mb) for each measured region of quadriceps femoris | 1 session constant-load bed-cycling + 1 interval bed-cycling session administered in 2 different days within 1 week.
  Differences between exercise protocols in oxygenated hemoglobin/myoglobin (OxyHb/Mb), deoxygenated hemoglobin/myoglobin (DeoxyHb/Mb) and total hemoglobin/myoglobin concentration (TotHb/Mb) for each measured region of quadriceps femoris (i.e., vastus lateralis, vastus medialis, rectus femoris upper part and rectus femoris lower part)
Differences in Median frequency of sEMG of different regions of quadriceps femoris | 1 session constant-load bed-cycling + 1 interval bed-cycling session administered in 2 different days within 1 week.
  Differences in Median frequency of sEMG of different regions of quadriceps femoris (i.e., vastus lateralis, vastus medialis, rectus femoris upper part and rectus femoris lower part) between exercise protocols
Differences in relative dispersion (RD) of sEMG values among the different regions of quadriceps femoris as indicator of heterogeneity of activation among different regions of quadriceps femoris muscle. | 1 session constant-load bed-cycling + 1 interval bed-cycling session administered in 2 different days within 1 week.
  Differences between exercise protocols in relative dispersion (RD) of sEMG values among the different regions of quadriceps femoris as indicator of heterogeneity of activation among different regions of quadriceps femoris muscle.
Differences between bed-cycling protocols in heart rate | constant-load and interval bed-cycling protocols administered in 2 different days within 1 week
  Assessed by monitoring vital signs
Differences between bed-cycling protocols in mean arterial blood pressure | constant-load and interval bed-cycling protocols administered in 2 different days within 1 week
  Assessed by monitoring vital signs
Differences between bed-cycling protocols in respiratory frequency | constant-load and interval bed-cycling protocols administered in 2 different days within 1 week
  Assessed by monitoring vital signs
Differences between bed-cycling protocols in minute ventilation | constant-load and interval bed-cycling protocols administered in 2 different days within 1 week
  In case of mechanically ventilated patients
Differences between bed-cycling protocols in tidal volume | constant-load and interval bed-cycling protocols administered in 2 different days within 1 week
  In case of mechanically ventilated patients
Differences between bed-cycling protocols in peripheral capillary oxygen saturation | constant-load and interval bed-cycling protocols administered in 2 different days within 1 week
  Assessed by monitoring vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Langer, Prof. Dr., Principal Investigator — KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium

REFERENCES:
- [Background] Anekwe DE, Biswas S, Bussieres A, Spahija J. Early rehabilitation reduces the likelihood of developing intensive care unit-acquired weakness: a systematic review and meta-analysis. Physiotherapy. 2020 Jun;107:1-10. doi: 10.1016/j.physio.2019.12.004. Epub 2019 Dec 19. PMID 32135387
- [Background] Clarissa C, Salisbury L, Rodgers S, Kean S. Early mobilisation in mechanically ventilated patients: a systematic integrative review of definitions and activities. J Intensive Care. 2019 Jan 17;7:3. doi: 10.1186/s40560-018-0355-z. eCollection 2019. PMID 30680218
- [Background] Supinski GS, Valentine EN, Netzel PF, Schroder EA, Wang L, Callahan LA. Does Standard Physical Therapy Increase Quadriceps Strength in Chronically Ventilated Patients? A Pilot Study. Crit Care Med. 2020 Nov;48(11):1595-1603. doi: 10.1097/CCM.0000000000004544. PMID 32826429
- [Background] Grunow JJ, Goll M, Carbon NM, Liebl ME, Weber-Carstens S, Wollersheim T. Differential contractile response of critically ill patients to neuromuscular electrical stimulation. Crit Care. 2019 Sep 10;23(1):308. doi: 10.1186/s13054-019-2540-4. PMID 31506074
- [Background] Reid JC, Clarke F, Cook DJ, Molloy A, Rudkowski JC, Stratford P, Kho ME. Feasibility, Reliability, Responsiveness, and Validity of the Patient-Reported Functional Scale for the Intensive Care Unit: A Pilot Study. J Intensive Care Med. 2020 Dec;35(12):1396-1404. doi: 10.1177/0885066618824534. Epub 2019 Jan 22. PMID 30669936
- [Background] Hoffman M, Clerckx B, Janssen K, Segers J, Demeyere I, Frickx B, Merckx E, Hermans G, Van der Meulen I, Van Lancker T, Ceulemans N, Van Hollebeke M, Langer D, Gosselink R. Early mobilization in clinical practice: the reliability and feasibility of the 'Start To Move' Protocol. Physiother Theory Pract. 2022 Jul;38(7):908-918. doi: 10.1080/09593985.2020.1805833. Epub 2020 Aug 31. PMID 32866055
- [Background] Nickels MR, Aitken LM, Barnett AG, Walsham J, McPhail SM. Acceptability, safety, and feasibility of in-bed cycling with critically ill patients. Aust Crit Care. 2020 May;33(3):236-243. doi: 10.1016/j.aucc.2020.02.007. Epub 2020 Apr 18. PMID 32317212